CLINICAL TRIAL: NCT06844227
Title: Perioperative Anticoagulant Use for Surgery Evaluation -Virtual Visit (PAUSE-Virtual), a Simple Perioperative Anticoagulant Management Approach, Replacing a Resource-intensive In-person Doctor-patient Consultation, With a Simple Virtual Care Model That Will Provide a New Standard of Care for Patients on a Direct Oral Anticoagulant or Warfarin and Require Elective Surgery/Procedure.
Brief Title: Perioperative Anticoagulant Use for Surgery Evaluation -Virtual Visit (PAUSE-Virtual)
Acronym: PAUSEVirtual
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: PAUSE Virtual (CTO 3854); 202104PJT-461879-CID-CEBA-5761 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-11-25; First posted 2025-02-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: anticoagulation; Atrial Fibrillation; Surgery; Oral Anticoagulant; Blood Thinner; DOAC; Interruption; Perioperative; Virtual; PAUSE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 mL whole blood sample, to be processed for plasma that will be frozen and stored at local sites until transfer to the Clinical Research Laboratory & Biobank at Hamilton Health Sciences, Hamilton, Ontario
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: warfarin-treated patients: Cohort 1: warfarin-treated patients with AF who receive virtual perioperative management
- Cohort 2: DOAC-treated patients: Cohort 2: DOAC-treated patients with AF who receive virtual perioperative management.
  Using this design, the investigator aims to show in Cohorts 1 and 2 that virtual management is non-inferior to benchmark in-person management, defined by 30-day postoperative rates of SSE ≤0.5% (with 95% confidence to exclude 1.5% rate) and MB ≤1.5% (with 95% confidence to exclude 3% rate).

SUMMARY:
The purpose of the PAUSE-Virtual Study is to show that by changing pre-surgery visits with patients taking a blood thinner (direct oral anticoagulant (apixaban, dabigatran, edoxaban, rivaroxaban or warfarin) when the participant requires elective surgery, using a standard, in-person proven approach, to a virtual visit, either telephone or video conference, is as safe. Patients who are receiving a blood thinner for the medical condition known as atrial fibrillation (AF) and require an elective surgery/procedure, is common. These patients have to stop taking their blood thinner for a certain time before the procedure to reduce serious complications of stroke or bleeding. For doctors who help manage these patients before a procedure, appointments have been traditionally done in-person. Patients receive instructions about when to stop and restart their blood thinners and taught how to self-administrator a short acting blood thinner (heparin) if needed. The COVID pandemic changed the way these appointments were done, making it important to contact these patients without them having to come to the hospital for an in person visit. Virtual patient care, by telephone or video conference, to communicate to patients about when to start and restart their blood thinner was necessary. This study wants to show that this virtual method of instruction, using a standardized plan of managing patient care, is easy, acceptable to patients and as safe when compared to an in-person meeting. Such instruction would also be cost-efficient standard post-pandemic. Prior work has shown that both a standard care of patients who are receiving blood thinners and a point-of-care decision "app", available through Thrombosis Canada (www.thrombosiscanada.ca) website, have been trusted during this virtual visit successfully. The investigator will show, by following up at 30 days, that this standardized management plan is safe and can be done virtually, with a low risk of stroke and major bleeding.

DETAILED DESCRIPTION:
The Clinical Problem: The management of patients who are taking warfarin or a direct oral anticoagulant (DOAC) and need an elective surgery/procedure is a common and important clinical problem: (i) ~200,000 patients/yr are assessed in Canada for such management and this will increase due to an ageing population and an increase in anticoagulant use; and (ii) if anticoagulants are not managed carefully, with evidence-based protocols, patients can be exposed to an increased risk for disabling stroke if anticoagulant interruption is too long or life-threatening bleeding if interruption is too short.

The Healthcare Delivery Problem: Perioperative management of anticoagulant therapy has been traditionally done in an in-person setting where patients receive instructions about when to stop and restart anticoagulants and, if needed, to receive teaching to self-administer heparin bridging. The COVID pandemic has upended this healthcare delivery model, necessitating virtual management by phone/video. Virtual patient care to manage perioperative anticoagulation has the potential to be an efficient and patient-friendly standard post-pandemic. However, to attain this objective, it must be reliably shown that virtually-administered, standardized, perioperative anticoagulation management is: (i) safe, with acceptably low rates of stroke and bleeding; (ii) easy to apply in practice; and (iii) acceptable to patients.

The foundation for this study is based on prior work by the investigator: (i) The investigator has led multicenter clinical trials (BRIDGE, PAUSE) that provide benchmarks for safe perioperative management of patients who are receiving warfarin or a DOAC; (ii) the management protocols from these trials were incorporated into a clinical decision tool that is available (cost-free) by Thrombosis Canada (www.thrombosiscanada.ca). This point-of-care app allows input of patient-specific information to manage individual patients with atrial fibrillation/flutter (AF) who are receiving warfarin or a DOAC and require an elective surgery/procedure. At the end of the assessment, a care-path summary is available as a PDF for clinicians and patients for downloading and printing.

The Opportunity: The pandemic has necessitated the adoption of virtual perioperative anticoagulant management but also has provided the opportunity to re-evaluate how such care can be safely delivered. Given that (i) perioperative anticoagulant interruption/resumption and heparin bridging protocols are standardized, and (ii) there is an easy-to-use, point-of-care, management app available, the investigator has a unique opportunity to apply evidence-informed protocols with user-friendly knowledge translation tools to assess the safety and acceptability to patients of virtual perioperative anticoagulant management.

The Solution: A prospective cohort study (non-RCT) assessing standardized virtual perioperative management in 2 cohorts of patients on warfarin or a DOAC who require an elective surgery/procedure.

Hypothesis & Postulates: (i) the investigator hypothesizes that virtual perioperative management will be safe for patient care, with 30-day postoperative rates of stroke/systemic embolism (SSE) ≤0.5% and major bleeding (MB) ≤1.5%. With a sample size of 847 patients in Cohort 1 and in Cohort 2, the investigator will have 90% power at the 95% level of significance to reject the null hypothesis that the observed rates are ≥1.5% for SSE and ≥3% for MB in each cohort. (ii) The investigator postulates (a) that virtual management will be as safe as in matched historical control groups who received benchmark in-person management, (b) that virtual management will reduce healthcare costs and costs to patients, and (c) that patients will be satisfied with virtual management and will be willing to receive this methods of healthcare delivery post-pandemic.

Significance: PAUSE-Virtual will shift perioperative anticoagulant management from a resource-intensive in-person model to a patient-friendly virtual model, establishing a standard-of-care option for 200,000 patients/yr in Canada. The investigator is a leading group in perioperative anticoagulant management worldwide, having done the landmark BRIDGE1 and PAUSE2 trials. There is no other research group (that the investigator knows of) that will do this trial, and it will not be funded by industry (no commercial interest).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older with AF/flutter (chronic, persistent, paroxysmal) that requires anticoagulation
* Receiving warfarin, with a target international normalized ratio (INR) range of 2.0-3.0, or a DOAC, comprising one of the following regimens: apixaban, 2.5 mg or 5 mg bid; edoxaban, 30 mg or 60 mg daily; dabigatran, 110 mg or 150 mg bid; or rivaroxaban, 15 mg or 20 mg daily
* Require an elective (planned, non-urgent) surgery or invasive medical or surgical procedure

Exclusion Criteria:

* Indication for anticoagulation is not AF/flutter (e.g., mechanical heart valve, VTE, other)
* Non-standard anticoagulant regimen used (e.g., warfarin INR 3-4, rivaroxaban 2.5 mg bid)
* In DOAC users only: creatinine clearance <25 mL/min (that preclude DOAC use)
* Cognitive impairment or psychiatric illness (that precludes reliable contact during follow-up)
* Unable or unwilling to provide consent for virtual care (in-person care will be provided)
* Previous participation in this study for an elective surgery/procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overall, the study population chosen is justified because: (i) AF/flutter is the dominant clinical indication for anticoagulant therapy; (ii) it is homogenous, thereby optimizing generalizability of study results; and (iii) it allows patient-level comparisons of outcomes with controls from the BRIDGE and PAUSE trials which included AF/flutter (but excluded patients with a MHV or VTE).
Sampling Method: Non-Probability Sample
Enrollment: 1780 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | From enrollment to end of 30 day follow up
  The investigator will determine 30-day post-procedure event rates with 95% confidence interval (CIs) for stroke/systemic embolism (SSE), major bleeding (MB) and, with a one-sided binomial test, will determine in Cohort 1 and Cohort 2 if the SSE rate is lower than 1.5%, and the MB rate is lower than 3%. The investigator will compare patient demographic (e.g., age, gender) and clinical characteristics (e.g., surgery type, SSE/MB risk) in Cohort 1 vs. Control 1 and Cohort 2 vs. Control 2 using Fisher's exact test, respectively, so as to compare SSE and MB in Cohorts and Controls, adjusting for key covariates (e.g., surgery type, anticoagulant type, gender) using multivariate logistic regression. The investigator will determine the proportions (and 95% CIs) for patient satisfaction categories in virtual care and willingness to receive future virtual care.

SECONDARY OUTCOMES:
Secondary Outcome 1 | From enrollment to end of 30 day follow up
  To demonstrate that virtual management is safe, as defined by 30-day postoperative rates of stroke/systemic embolism (SSE) of ≤0.5% and major bleeding (MB) of ≤1.5% with ability to exclude rates of SSE and MB of 1.5% and 3.0%, with a sample of 847 patients in Cohorts 1 and 2, the investigator will have 90% power at the 95% level of significance to reject the null hypothesis that the observed rate of SSE is ≥1.5% and MB is ≥3.0%. This sample size of 847 is increased by 5% to 890 patients per Cohort (1,780 total) to account for cancelled surgeries/procedures and patients lost to follow-up.
Secondary Outcome 2 | From enrollment to end of 30 day follow up
  The investigator will determine the cost effectiveness of the virtual management compared with in-person care from both public payer and societal perspectives. Health resource use will be collected alongside the clinical data collection that includes physician, nursing and pharmacist consultation time, medication, diagnostics and procedures, and hospitalization. Patient's time and travel costs will also be included in the analysis from the societal perspective. Incremental cost effectiveness ratio between each of the cohort and corresponding control group will be calculated. 95% confidence interval of the ratio will be estimated using non-parametric bootstrapping approach. Cost effectiveness acceptability curves will be used to show the probability of virtual care being cost effective compared with in person care over a wide range of willingness-to-pay values.

CONTACTS AND LOCATIONS:
Overall Officials: James D Douketis, MD, Principal Investigator — McMaster University/St. Joseph's Healthcare
Locations (10):
- United States (4):
  - Endeavor Health - Northshore, Evanston, Illinois
  - Henry Ford, Detroit, Michigan
  - Northwell Health, Great Neck, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Canada (5):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joesph's Healthcare, Hamilton, Ontario
  - Juravinski, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
- Larissa University Hospital, Larissa, Larisa, Greece

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared. All data reported as part of the study is aggregate data.

REFERENCES:
- [Background] Jamula E, Woods K, Verhovsek M, Douketis JD, McDonald E. Comparison of pain and ecchymosis with low-molecular-weight heparin vs. unfractionated heparin in patients requiring bridging anticoagulation after warfarin interruption: a randomized trial. J Thromb Thrombolysis. 2009 Oct;28(3):266-8. doi: 10.1007/s11239-009-0312-8. Epub 2009 Feb 14. PMID 19219405
- [Background] Brown SD, Lee K, Schoffman DE, King AC, Crawley LM, Kiernan M. Minority recruitment into clinical trials: experimental findings and practical implications. Contemp Clin Trials. 2012 Jul;33(4):620-3. doi: 10.1016/j.cct.2012.03.003. Epub 2012 Mar 16. PMID 22449836
- [Background] Clark LT, Watkins L, Pina IL, Elmer M, Akinboboye O, Gorham M, Jamerson B, McCullough C, Pierre C, Polis AB, Puckrein G, Regnante JM. Increasing Diversity in Clinical Trials: Overcoming Critical Barriers. Curr Probl Cardiol. 2019 May;44(5):148-172. doi: 10.1016/j.cpcardiol.2018.11.002. Epub 2018 Nov 9. PMID 30545650
- [Background] Amorrortu RP, Arevalo M, Vernon SW, Mainous AG 3rd, Diaz V, McKee MD, Ford ME, Tilley BC. Recruitment of racial and ethnic minorities to clinical trials conducted within specialty clinics: an intervention mapping approach. Trials. 2018 Feb 17;19(1):115. doi: 10.1186/s13063-018-2507-9. PMID 29454389
- [Background] Shaw JR, Zhang T, Le Gal G, Douketis J, Carrier M. Perioperative interruption of direct oral anticoagulants and vitamin K antagonists in patients with atrial fibrillation: A comparative analysis. Res Pract Thromb Haemost. 2020 Jan 20;4(1):131-140. doi: 10.1002/rth2.12285. eCollection 2020 Jan. PMID 31989095
- [Background] Skeith L, Taylor J, Lazo-Langner A, Kovacs MJ. Conservative perioperative anticoagulation management in patients with chronic venous thromboembolic disease: a cohort study. J Thromb Haemost. 2012 Nov;10(11):2298-304. doi: 10.1111/j.1538-7836.2012.04907.x. PMID 22925003
- [Background] Cahill TJ, Chen M, Hayashida K, Latib A, Modine T, Piazza N, Redwood S, Sondergaard L, Prendergast BD. Transcatheter aortic valve implantation: current status and future perspectives. Eur Heart J. 2018 Jul 21;39(28):2625-2634. doi: 10.1093/eurheartj/ehy244. PMID 29718148
- [Background] Isaacs AJ, Shuhaiber J, Salemi A, Isom OW, Sedrakyan A. National trends in utilization and in-hospital outcomes of mechanical versus bioprosthetic aortic valve replacements. J Thorac Cardiovasc Surg. 2015 May;149(5):1262-9.e3. doi: 10.1016/j.jtcvs.2015.01.052. Epub 2015 Feb 11. PMID 25791947
- [Background] Andrade JG, Aguilar M, Atzema C, Bell A, Cairns JA, Cheung CC, Cox JL, Dorian P, Gladstone DJ, Healey JS, Khairy P, Leblanc K, McMurtry MS, Mitchell LB, Nair GM, Nattel S, Parkash R, Pilote L, Sandhu RK, Sarrazin JF, Sharma M, Skanes AC, Talajic M, Tsang TSM, Verma A, Verma S, Whitlock R, Wyse DG, Macle L; Members of the Secondary Panel. The 2020 Canadian Cardiovascular Society/Canadian Heart Rhythm Society Comprehensive Guidelines for the Management of Atrial Fibrillation. Can J Cardiol. 2020 Dec;36(12):1847-1948. doi: 10.1016/j.cjca.2020.09.001. Epub 2020 Oct 22. PMID 33191198
- [Background] Andersson T, Magnuson A, Bryngelsson IL, Frobert O, Henriksson KM, Edvardsson N, Poci D. Gender-related differences in risk of cardiovascular morbidity and all-cause mortality in patients hospitalized with incident atrial fibrillation without concomitant diseases: a nationwide cohort study of 9519 patients. Int J Cardiol. 2014 Nov 15;177(1):91-9. doi: 10.1016/j.ijcard.2014.09.092. Epub 2014 Oct 11. PMID 25499348
- [Background] Pancholy SB, Sharma PS, Pancholy DS, Patel TM, Callans DJ, Marchlinski FE. Meta-analysis of gender differences in residual stroke risk and major bleeding in patients with nonvalvular atrial fibrillation treated with oral anticoagulants. Am J Cardiol. 2014 Feb 1;113(3):485-90. doi: 10.1016/j.amjcard.2013.10.035. Epub 2013 Nov 11. PMID 24315113
- [Background] McAlister FA, Garrison S, Kosowan L, Ezekowitz JA, Singer A. Use of Direct Oral Anticoagulants in Canadian Primary Care Practice 2010-2015: A Cohort Study From the Canadian Primary Care Sentinel Surveillance Network. J Am Heart Assoc. 2018 Jan 26;7(3):e007603. doi: 10.1161/JAHA.117.007603. PMID 29374047
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Czeisler ME, Marynak K, Clarke KEN, Salah Z, Shakya I, Thierry JM, Ali N, McMillan H, Wiley JF, Weaver MD, Czeisler CA, Rajaratnam SMW, Howard ME. Delay or Avoidance of Medical Care Because of COVID-19-Related Concerns - United States, June 2020. MMWR Morb Mortal Wkly Rep. 2020 Sep 11;69(36):1250-1257. doi: 10.15585/mmwr.mm6936a4. PMID 32915166
- [Background] Woolf SH, Chapman DA, Sabo RT, Weinberger DM, Hill L. Excess Deaths From COVID-19 and Other Causes, March-April 2020. JAMA. 2020 Aug 4;324(5):510-513. doi: 10.1001/jama.2020.11787. PMID 32609307
- [Background] Weinberger DM, Chen J, Cohen T, Crawford FW, Mostashari F, Olson D, Pitzer VE, Reich NG, Russi M, Simonsen L, Watkins A, Viboud C. Estimation of Excess Deaths Associated With the COVID-19 Pandemic in the United States, March to May 2020. JAMA Intern Med. 2020 Oct 1;180(10):1336-1344. doi: 10.1001/jamainternmed.2020.3391. PMID 32609310
- [Background] Sackett DL. Bias in analytic research. J Chronic Dis. 1979;32(1-2):51-63. doi: 10.1016/0021-9681(79)90012-2. No abstract available. PMID 447779
- [Background] Spyropoulos AC, Myrka A, Triller DM, Ragan S, York C, King JM, Lee TK. Uptake and Utilization of the Management of Anticoagulation in the Periprocedural Period App: Longitudinal Analysis. JMIR Mhealth Uhealth. 2018 Dec 21;6(12):e11090. doi: 10.2196/11090. PMID 30578235
- [Background] Spyropoulos AC, Giannis D, Cohen J, John S, Myrka A, Inlall D, Qiu M, Akgul S, Hyman RJ, Wang JJ. Implementation of the Management of Anticoagulation in the Periprocedural Period App Into an Electronic Health Record: A Prospective Cohort Study. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620925910. doi: 10.1177/1076029620925910. PMID 32633538
- [Background] Sherwood MW, Douketis JD, Patel MR, Piccini JP, Hellkamp AS, Lokhnygina Y, Spyropoulos AC, Hankey GJ, Singer DE, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Becker RC; ROCKET AF Investigators. Outcomes of temporary interruption of rivaroxaban compared with warfarin in patients with nonvalvular atrial fibrillation: results from the rivaroxaban once daily, oral, direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and embolism trial in atrial fibrillation (ROCKET AF). Circulation. 2014 May 6;129(18):1850-9. doi: 10.1161/CIRCULATIONAHA.113.005754. Epub 2014 Feb 19. PMID 24552831
- [Background] Spyropoulos AC, Douketis JD. Guidelines for antithrombotic therapy: periprocedural management of antithrombotic therapy and use of bridging anticoagulation. Int Angiol. 2008 Aug;27(4):333-43. No abstract available. PMID 18677297
- [Background] Spyropoulos AC, Albaladejo P, Godier A, Greinacher A, Hron G, Levy JH, Samama CM, Douketis JD. Periprocedural antiplatelet therapy: recommendations for standardized reporting in patients on antiplatelet therapy: communication from the SSC of the ISTH. J Thromb Haemost. 2013 Aug;11(8):1593-6. doi: 10.1111/jth.12282. No abstract available. PMID 23647986
- [Background] Spyropoulos AC, Brohi K, Caprini J, Samama CM, Siegal D, Tafur A, Verhamme P, Douketis JD; SSC Subcommittee on Perioperative and Critical Care Thrombosis and Haemostasis of the International Society on Thrombosis and Haemostasis. Scientific and Standardization Committee Communication: Guidance document on the periprocedural management of patients on chronic oral anticoagulant therapy: Recommendations for standardized reporting of procedural/surgical bleed risk and patient-specific thromboembolic risk. J Thromb Haemost. 2019 Nov;17(11):1966-1972. doi: 10.1111/jth.14598. Epub 2019 Aug 22. No abstract available. PMID 31436045
- [Background] Spyropoulos AC, Douketis JD, Gerotziafas G, Kaatz S, Ortel TL, Schulman S; Subcommittee on Control of Anticoagulation of the SSC of the ISTH. Periprocedural antithrombotic and bridging therapy: recommendations for standardized reporting in patients with arterial indications for chronic oral anticoagulant therapy. J Thromb Haemost. 2012 Apr;10(4):692-4. doi: 10.1111/j.1538-7836.2012.04630.x. No abstract available. PMID 22934291
- [Background] Douketis JD, Berger PB, Dunn AS, Jaffer AK, Spyropoulos AC, Becker RC, Ansell J. The perioperative management of antithrombotic therapy: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):299S-339S. doi: 10.1378/chest.08-0675. PMID 18574269
- [Background] Clark NP, Douketis JD, Hasselblad V, Schulman S, Kindzelski AL, Ortel TL; BRIDGE Investigators. Predictors of perioperative major bleeding in patients who interrupt warfarin for an elective surgery or procedure: Analysis of the BRIDGE trial. Am Heart J. 2018 Jan;195:108-114. doi: 10.1016/j.ahj.2017.09.015. Epub 2017 Sep 21. PMID 29224638
- [Background] Kaatz S, Douketis JD, Zhou H, Gage BF, White RH. Risk of stroke after surgery in patients with and without chronic atrial fibrillation. J Thromb Haemost. 2010 May;8(5):884-90. doi: 10.1111/j.1538-7836.2010.03781.x. Epub 2010 Jan 24. PMID 20096001
- [Background] MacDougall K, Douketis JD, Li N, Clark NP, Tafur A, D'Astous J, Duncan J, Schulman S, Spyropoulos AC. Effect of Direct Oral Anticoagulant, Patient, and Surgery Characteristics on Clinical Outcomes in the Perioperative Anticoagulation Use for Surgery Evaluation Study. TH Open. 2020 Sep 23;4(3):e255-e262. doi: 10.1055/s-0040-1716512. eCollection 2020 Jul. PMID 32984757
- [Background] Tafur AJ, Clark NP, Spyropoulos AC, Li N, Kaplovitch E, MacDougall K, Schulman S, Caprini JA, Douketis J. Predictors of Bleeding in the Perioperative Anticoagulant Use for Surgery Evaluation Study. J Am Heart Assoc. 2020 Oct 20;9(19):e017316. doi: 10.1161/JAHA.120.017316. Epub 2020 Sep 24. PMID 32969288
- [Background] Shaw JR, Li N, Vanassche T, Coppens M, Spyropoulos AC, Syed S, Radwi M, Duncan J, Schulman S, Douketis JD. Predictors of preprocedural direct oral anticoagulant levels in patients having an elective surgery or procedure. Blood Adv. 2020 Aug 11;4(15):3520-3527. doi: 10.1182/bloodadvances.2020002335. PMID 32756938
- [Background] Douketis JD, Syed S, Schulman S. Periprocedural Management of Direct Oral Anticoagulants: Comment on the 2015 American Society of Regional Anesthesia and Pain Medicine Guidelines. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):127-9. doi: 10.1097/AAP.0000000000000360. No abstract available. PMID 26882272
- [Background] Kim PY, Di Giuseppantonio LR, Wu C, Douketis JD, Gross PL. An assay to measure levels of factor Xa inhibitors in blood and plasma. J Thromb Haemost. 2019 Jul;17(7):1153-1159. doi: 10.1111/jth.14451. Epub 2019 May 10. PMID 30985986
- [Background] Dube C, Douketis JD, Moffat KA, Schulman S, Blais N. Basic coagulation tests as surrogates of dabigatran levels in a pre-operative setting: Analysis of five activated partial thromboplastin time reagents and thrombin time. Thromb Res. 2018 Nov;171:62-67. doi: 10.1016/j.thromres.2018.09.051. Epub 2018 Sep 19. PMID 30261356
- [Background] Douketis J, Schulman S, Syed S. Reply to Dr Lessire et al. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):788. doi: 10.1097/AAP.0000000000000478. No abstract available. PMID 27662066
- [Background] Douketis JD, Johnson JA, Turpie AG. Low-molecular-weight heparin as bridging anticoagulation during interruption of warfarin: assessment of a standardized periprocedural anticoagulation regimen. Arch Intern Med. 2004 Jun 28;164(12):1319-26. doi: 10.1001/archinte.164.12.1319. PMID 15226166
- [Background] Schulman S, Carrier M, Lee AY, Shivakumar S, Blostein M, Spencer FA, Solymoss S, Barty R, Wang G, Heddle N, Douketis JD; Periop Dabigatran Study Group. Perioperative Management of Dabigatran: A Prospective Cohort Study. Circulation. 2015 Jul 21;132(3):167-73. doi: 10.1161/CIRCULATIONAHA.115.015688. Epub 2015 May 12. PMID 25966905
- [Background] Douketis JD, Murphy SA, Antman EM, Grip LT, Mercuri MF, Ruff CT, Weitz JI, Braunwald E, Giugliano RP. Peri-operative Adverse Outcomes in Patients with Atrial Fibrillation Taking Warfarin or Edoxaban: Analysis of the ENGAGE AF-TIMI 48 Trial. Thromb Haemost. 2018 Jun;118(6):1001-1008. doi: 10.1055/s-0038-1645856. Epub 2018 May 3. PMID 29723874
- [Background] Douketis J, Wang J, Cuddy K, Wagler M, Kinnon K, Crowther M. The safety of co-administered continuous epidural analgesia and low-molecular-weight heparin after major orthopedic surgery: assessment of a standardized patient management protocol. Thromb Haemost. 2006 Sep;96(3):387-9. doi: 10.1160/TH06-06-0303. No abstract available. PMID 16953285
- [Background] Douketis JD, Wang G, Chan N, Eikelboom JW, Syed S, Barty R, Moffat KA, Spencer FA, Blostein M, Schulman S. Effect of standardized perioperative dabigatran interruption on the residual anticoagulation effect at the time of surgery or procedure. J Thromb Haemost. 2016 Jan;14(1):89-97. doi: 10.1111/jth.13178. Epub 2016 Jan 4. PMID 26512880
- [Background] Douketis JD, Healey JS, Brueckmann M, Fraessdorf M, Spyropoulos AC, Wallentin L, Oldgren J, Reilly P, Ezekowitz MD, Connolly SJ, Yusuf S, Eikelboom JW. Urgent surgery or procedures in patients taking dabigatran or warfarin: Analysis of perioperative outcomes from the RE-LY trial. Thromb Res. 2016 Mar;139:77-81. doi: 10.1016/j.thromres.2016.01.004. Epub 2016 Jan 9. PMID 26916299
- [Background] Douketis JD, Healey JS, Brueckmann M, Eikelboom JW, Ezekowitz MD, Fraessdorf M, Noack H, Oldgren J, Reilly P, Spyropoulos AC, Wallentin L, Connolly SJ. Perioperative bridging anticoagulation during dabigatran or warfarin interruption among patients who had an elective surgery or procedure. Substudy of the RE-LY trial. Thromb Haemost. 2015 Mar;113(3):625-32. doi: 10.1160/TH14-04-0305. Epub 2014 Dec 4. PMID 25472710
- [Background] Spyropoulos AC, Turpie AG, Dunn AS, Kaatz S, Douketis J, Jacobson A, Petersen H; REGIMEN Investigators. Perioperative bridging therapy with unfractionated heparin or low-molecular-weight heparin in patients with mechanical prosthetic heart valves on long-term oral anticoagulants (from the REGIMEN Registry). Am J Cardiol. 2008 Oct 1;102(7):883-9. doi: 10.1016/j.amjcard.2008.05.042. Epub 2008 Jul 31. PMID 18805116
- [Background] Bell BR, Spyropoulos AC, Douketis JD. Perioperative Management of the Direct Oral Anticoagulants: A Case-Based Review. Hematol Oncol Clin North Am. 2016 Oct;30(5):1073-84. doi: 10.1016/j.hoc.2016.05.005. PMID 27637308
- [Background] Shaw JR, Kaplovitch E, Douketis J. Periprocedural Management of Oral Anticoagulation. Med Clin North Am. 2020 Jul;104(4):709-726. doi: 10.1016/j.mcna.2020.02.005. Epub 2020 May 12. PMID 32505262
- [Background] Douketis JD. Perioperative management of warfarin therapy: to bridge or not to bridge, that is the question. Mayo Clin Proc. 2008 Jun;83(6):628-9. doi: 10.4065/83.6.628. No abstract available. PMID 18533078
- [Background] Spyropoulos AC. Bridging therapy and oral anticoagulation: current and future prospects. Curr Opin Hematol. 2010 Sep;17(5):444-9. doi: 10.1097/MOH.0b013e32833c077b. PMID 20613508
- [Background] Spyropoulos AC. Perioperative bridging therapy for the at-risk patient on chronic anticoagulation. Dis Mon. 2005 Feb-Mar;51(2-3):183-93. doi: 10.1016/j.disamonth.2005.03.014. No abstract available. PMID 15900271
- [Background] Spyropoulos AC. Bridging of oral anticoagulation therapy for invasive procedures. Curr Hematol Rep. 2005 Sep;4(5):405-13. PMID 16131443
- [Background] Douketis JD, Crowther MA, Cherian SS, Kearon CB. Physician preferences for perioperative anticoagulation in patients with a mechanical heart valve who are undergoing elective noncardiac surgery. Chest. 1999 Nov;116(5):1240-6. doi: 10.1378/chest.116.5.1240. PMID 10559081
- [Background] Douketis JD, Crowther MA, Cherian SS. Perioperative anticoagulation in patients with chronic atrial fibrillation who are undergoing elective surgery: results of a physician survey. Can J Cardiol. 2000 Mar;16(3):326-30. PMID 10744795
- [Background] Douketis JD, Bakhsh E. Perioperative management of antithrombotic therapy. Pol Arch Med Wewn. 2008 Apr;118(4):201-8. PMID 18575419
- [Background] Douketis JD. Pharmacologic properties of the new oral anticoagulants: a clinician-oriented review with a focus on perioperative management. Curr Pharm Des. 2010;16(31):3436-41. doi: 10.2174/138161210793563338. PMID 20858185
- [Background] Douketis J, Bell AD, Eikelboom J, Liew A. Approach to the new oral anticoagulants in family practice: part 2: addressing frequently asked questions. Can Fam Physician. 2014 Nov;60(11):997-1001. PMID 25392439
- [Background] Douketis JD. Perioperative anticoagulation management in patients who are receiving oral anticoagulant therapy: a practical guide for clinicians. Thromb Res. 2002 Oct 1;108(1):3-13. doi: 10.1016/s0049-3848(02)00387-0. PMID 12586125
- [Background] Douketis J, Cervi A. Managing patients who are receiving warfarin or a direct oral anticoagulant and need an elective surgery or procedure. Blood Adv. 2019 Jun 25;3(12):1925. doi: 10.1182/bloodadvances.2019000171. No abstract available. PMID 31239247
- [Background] Jamula E, Lloyd NS, Schwalm JD, Airaksinen KE, Douketis JD. Safety of uninterrupted anticoagulation in patients requiring elective coronary angiography with or without percutaneous coronary intervention: a systematic review and metaanalysis. Chest. 2010 Oct;138(4):840-7. doi: 10.1378/chest.09-2603. Epub 2010 Apr 30. PMID 20435662
- [Background] Jamula E, Anderson J, Douketis JD. Safety of continuing warfarin therapy during cataract surgery: a systematic review and meta-analysis. Thromb Res. 2009 Jul;124(3):292-9. doi: 10.1016/j.thromres.2009.01.007. Epub 2009 Feb 23. PMID 19233450
- [Background] Shaw JR, Woodfine JD, Douketis J, Schulman S, Carrier M. Perioperative interruption of direct oral anticoagulants in patients with atrial fibrillation: A systematic review and meta-analysis. Res Pract Thromb Haemost. 2018 Feb 16;2(2):282-290. doi: 10.1002/rth2.12076. eCollection 2018 Apr. PMID 30046730
- [Background] Siegal D, Yudin J, Kaatz S, Douketis JD, Lim W, Spyropoulos AC. Periprocedural heparin bridging in patients receiving vitamin K antagonists: systematic review and meta-analysis of bleeding and thromboembolic rates. Circulation. 2012 Sep 25;126(13):1630-9. doi: 10.1161/CIRCULATIONAHA.112.105221. Epub 2012 Aug 21. PMID 22912386
- [Background] Asiri A, AlBishi S, AlMadani W, ElMetwally A, Househ M. The Use of Telemedicine in Surgical Care: a Systematic Review. Acta Inform Med. 2018 Oct;26(3):201-206. doi: 10.5455/aim.2018.26.201-206. PMID 30515013
- [Background] Lesher AP, Shah SR. Telemedicine in the perioperative experience. Semin Pediatr Surg. 2018 Apr;27(2):102-106. doi: 10.1053/j.sempedsurg.2018.02.007. Epub 2018 Feb 7. PMID 29548350
- [Background] Brundisini F, Giacomini M, DeJean D, Vanstone M, Winsor S, Smith A. Chronic disease patients' experiences with accessing health care in rural and remote areas: a systematic review and qualitative meta-synthesis. Ont Health Technol Assess Ser. 2013 Sep 1;13(15):1-33. eCollection 2013. PMID 24228078
- [Background] Cevik M, Bamford CGG, Ho A. COVID-19 pandemic-a focused review for clinicians. Clin Microbiol Infect. 2020 Jul;26(7):842-847. doi: 10.1016/j.cmi.2020.04.023. Epub 2020 Apr 25. PMID 32344166
- [Background] COVIDSurg Collaborative. Global guidance for surgical care during the COVID-19 pandemic. Br J Surg. 2020 Aug;107(9):1097-1103. doi: 10.1002/bjs.11646. Epub 2020 Apr 15. PMID 32293715
- [Background] COVIDSurg Collaborative. Elective surgery cancellations due to the COVID-19 pandemic: global predictive modelling to inform surgical recovery plans. Br J Surg. 2020 Oct;107(11):1440-1449. doi: 10.1002/bjs.11746. Epub 2020 Jun 13. PMID 32395848
- [Background] Holman N, Knighton P, Kar P, O'Keefe J, Curley M, Weaver A, Barron E, Bakhai C, Khunti K, Wareham NJ, Sattar N, Young B, Valabhji J. Risk factors for COVID-19-related mortality in people with type 1 and type 2 diabetes in England: a population-based cohort study. Lancet Diabetes Endocrinol. 2020 Oct;8(10):823-833. doi: 10.1016/S2213-8587(20)30271-0. Epub 2020 Aug 13. PMID 32798471
- [Background] Jordan RE, Adab P, Cheng KK. Covid-19: risk factors for severe disease and death. BMJ. 2020 Mar 26;368:m1198. doi: 10.1136/bmj.m1198. No abstract available. PMID 32217618
- [Background] Mihalj M, Carrel T, Gregoric ID, Andereggen L, Zinn PO, Doll D, Stueber F, Gabriel RA, Urman RD, Luedi MM. Telemedicine for preoperative assessment during a COVID-19 pandemic: Recommendations for clinical care. Best Pract Res Clin Anaesthesiol. 2020 Jun;34(2):345-351. doi: 10.1016/j.bpa.2020.05.001. Epub 2020 May 14. PMID 32711839
- [Background] Miner H, Fatehi A, Ring D, Reichenberg JS. Clinician Telemedicine Perceptions During the COVID-19 Pandemic. Telemed J E Health. 2021 May;27(5):508-512. doi: 10.1089/tmj.2020.0295. Epub 2020 Sep 18. PMID 32946364
- [Background] Douketis JD, Syed S, Li N, Narouze S, Radwi M, Duncan J, Schulman S, Spyropoulos AC. A physician survey of perioperative neuraxial anesthesia management in patients on a direct oral anticoagulant. Res Pract Thromb Haemost. 2020 Dec 16;5(1):159-167. doi: 10.1002/rth2.12430. eCollection 2021 Jan. PMID 33537540
- [Background] Spencer NH, Sardo LA, Cordell JP, Douketis JD. Structure and function of a perioperative anticoagulation management clinic. Thromb Res. 2019 Oct;182:167-174. doi: 10.1016/j.thromres.2019.08.007. Epub 2019 Aug 23. PMID 31494438
- [Background] Spyropoulos AC, Douketis JD. How I treat anticoagulated patients undergoing an elective procedure or surgery. Blood. 2012 Oct 11;120(15):2954-62. doi: 10.1182/blood-2012-06-415943. Epub 2012 Aug 28. PMID 22932800
- [Background] Spyropoulos AC, Bauersachs RM, Omran H, Cohen M. Periprocedural bridging therapy in patients receiving chronic oral anticoagulation therapy. Curr Med Res Opin. 2006 Jun;22(6):1109-22. doi: 10.1185/030079906X104858. PMID 16846544
- [Background] Douketis JD. Perioperative management of patients who are receiving warfarin therapy: an evidence-based and practical approach. Blood. 2011 May 12;117(19):5044-9. doi: 10.1182/blood-2011-02-329979. Epub 2011 Mar 17. No abstract available. PMID 21415266
- [Background] Douketis JD. Perioperative management of patients receiving anticoagulant or antiplatelet therapy: a clinician-oriented and practical approach. Hosp Pract (1995). 2011 Oct;39(4):41-54. doi: 10.3810/hp.2011.10.921. PMID 22056822
- [Background] Steinberg BA, Hellkamp AS, Lokhnygina Y, Halperin JL, Breithardt G, Passman R, Hankey GJ, Patel MR, Becker RC, Singer DE, Hacke W, Berkowitz SD, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Piccini JP; ROCKET AF Steering Committee and Investigators. Use and outcomes of antiarrhythmic therapy in patients with atrial fibrillation receiving oral anticoagulation: results from the ROCKET AF trial. Heart Rhythm. 2014 Jun;11(6):925-32. doi: 10.1016/j.hrthm.2014.03.006. Epub 2014 May 13. PMID 24833235
- [Background] Broderick JP, Bonomo JB, Kissela BM, Khoury JC, Moomaw CJ, Alwell K, Woo D, Flaherty ML, Khatri P, Adeoye O, Ferioli S, Kleindorfer DO. Withdrawal of antithrombotic agents and its impact on ischemic stroke occurrence. Stroke. 2011 Sep;42(9):2509-14. doi: 10.1161/STROKEAHA.110.611905. Epub 2011 Jun 30. PMID 21719769
- [Background] Spyropoulos AC, Al-Badri A, Sherwood MW, Douketis JD. Periprocedural management of patients receiving a vitamin K antagonist or a direct oral anticoagulant requiring an elective procedure or surgery. J Thromb Haemost. 2016 May;14(5):875-85. doi: 10.1111/jth.13305. Epub 2016 Apr 7. PMID 26988871
- [Background] Barnes GD, Lucas E, Alexander GC, Goldberger ZD. National Trends in Ambulatory Oral Anticoagulant Use. Am J Med. 2015 Dec;128(12):1300-5.e2. doi: 10.1016/j.amjmed.2015.05.044. Epub 2015 Jul 2. PMID 26144101
- [Background] Weitz JI, Semchuk W, Turpie AG, Fisher WD, Kong C, Ciaccia A, Cairns JA. Trends in Prescribing Oral Anticoagulants in Canada, 2008-2014. Clin Ther. 2015 Nov 1;37(11):2506-2514.e4. doi: 10.1016/j.clinthera.2015.09.008. Epub 2015 Oct 16. PMID 26481493
- [Background] Gao L, Tadrous M, Knowles S, Mamdani M, Paterson JM, Juurlink D, Gomes T. Prior Authorization and Canadian Public Utilization of Direct-Acting Oral Anticoagulants. Healthc Policy. 2017 Nov;13(2):68-78. doi: 10.12927/hcpol.2017.25321. PMID 29274228
- [Background] Healey JS, Eikelboom J, Douketis J, Wallentin L, Oldgren J, Yang S, Themeles E, Heidbuchel H, Avezum A, Reilly P, Connolly SJ, Yusuf S, Ezekowitz M; RE-LY Investigators. Periprocedural bleeding and thromboembolic events with dabigatran compared with warfarin: results from the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) randomized trial. Circulation. 2012 Jul 17;126(3):343-8. doi: 10.1161/CIRCULATIONAHA.111.090464. Epub 2012 Jun 14. PMID 22700854
- [Background] Douketis JD, Spyropoulos AC, Spencer FA, Mayr M, Jaffer AK, Eckman MH, Dunn AS, Kunz R. Perioperative management of antithrombotic therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e326S-e350S. doi: 10.1378/chest.11-2298. PMID 22315266
- [Background] Proietti M, Laroche C, Opolski G, Maggioni AP, Boriani G, Lip GYH; AF Gen Pilot Investigators. 'Real-world' atrial fibrillation management in Europe: observations from the 2-year follow-up of the EURObservational Research Programme-Atrial Fibrillation General Registry Pilot Phase. Europace. 2017 May 1;19(5):722-733. doi: 10.1093/europace/euw112. PMID 27194538
- [Background] Steinberg BA, Gao H, Shrader P, Pieper K, Thomas L, Camm AJ, Ezekowitz MD, Fonarow GC, Gersh BJ, Goldhaber S, Haas S, Hacke W, Kowey PR, Ansell J, Mahaffey KW, Naccarelli G, Reiffel JA, Turpie A, Verheugt F, Piccini JP, Kakkar A, Peterson ED, Fox KAA; GARFIELD-AF; ORBIT-AF Investigators. International trends in clinical characteristics and oral anticoagulation treatment for patients with atrial fibrillation: Results from the GARFIELD-AF, ORBIT-AF I, and ORBIT-AF II registries. Am Heart J. 2017 Dec;194:132-140. doi: 10.1016/j.ahj.2017.08.011. Epub 2017 Aug 24. PMID 29223431
- [Background] Williams BA, Honushefsky AM, Berger PB. Temporal Trends in the Incidence, Prevalence, and Survival of Patients With Atrial Fibrillation From 2004 to 2016. Am J Cardiol. 2017 Dec 1;120(11):1961-1965. doi: 10.1016/j.amjcard.2017.08.014. Epub 2017 Aug 30. PMID 29033050
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Douketis JD, Spyropoulos AC, Duncan J, Carrier M, Le Gal G, Tafur AJ, Vanassche T, Verhamme P, Shivakumar S, Gross PL, Lee AYY, Yeo E, Solymoss S, Kassis J, Le Templier G, Kowalski S, Blostein M, Shah V, MacKay E, Wu C, Clark NP, Bates SM, Spencer FA, Arnaoutoglou E, Coppens M, Arnold DM, Caprini JA, Li N, Moffat KA, Syed S, Schulman S. Perioperative Management of Patients With Atrial Fibrillation Receiving a Direct Oral Anticoagulant. JAMA Intern Med. 2019 Nov 1;179(11):1469-1478. doi: 10.1001/jamainternmed.2019.2431. PMID 31380891
- [Background] Douketis JD, Spyropoulos AC, Kaatz S, Becker RC, Caprini JA, Dunn AS, Garcia DA, Jacobson A, Jaffer AK, Kong DF, Schulman S, Turpie AG, Hasselblad V, Ortel TL; BRIDGE Investigators. Perioperative Bridging Anticoagulation in Patients with Atrial Fibrillation. N Engl J Med. 2015 Aug 27;373(9):823-33. doi: 10.1056/NEJMoa1501035. Epub 2015 Jun 22. PMID 26095867
- See also: Valentine D GM, Grissinger M. . Valentine D, Gaunt MJ, Grissinger M. Identifying Patient Harm from Direct Oral Anticoagulants. Available from http://patientsafety.pa.gov/ADVISORIES/Pages/201806_DOACs.aspx. 2020 — http://patientsafety.pa.gov/ADVISORIES/Pages/201806_DOACs.aspx